CLINICAL TRIAL: NCT05106062
Title: Economic and Clinical Benefit of Remote Monitoring Among Defibrillator Patients by Indication Subgroups (BENEFIT-RM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2020-0075
Record Dates: First submitted 2021-10-05; First posted 2021-11-03 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Patients With Defibrillator
Keywords: defibrillator; remote monitoring; benefit; economic; clinical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Monitoring follow up (Experimental): This group will turn on the RM function 0 to 45 days after defibrillator implantation. Patient should be seen at clinic once a year, or if there is any adverse event notification
  Interventions: Device: on remote monitoring
- Conventional Follow up (No Intervention): This group will not turn on remote monitoring function of defibrillator. Patient should be seen at clinic according to center's custom but no longer than 6 months between each visit

INTERVENTIONS:
Device: on remote monitoring — This group will turn on the RM function 0 to 45 days after defibrillator implantation. Patient should be seen at clinic once a year, or if there is any adverse event notification
  Arms: Remote Monitoring follow up

SUMMARY:
Remote monitoring is now universally available for all cardiac implantable electronic devices (CIEDs), and it has become the standard of care for the management of patients with these devices. In many countries, it is being proven that patients with implantable defibrillator (ICD) or cardiac resynchronizing therapy (CRT) can benefit from remote monitoring (RM) both economically and clinically. From previous RM related clinical studies, it is reasonably accepted that hospitalization cost and mortality rate is comparably higher in defibrillator patients compared to pacemaker indicated patients.

However, it is yet to be discovered which group of defibrillator patients are the most beneficiaries using remote monitoring system. In this study, the investigators would further categorize defibrillator patients into different indication subgroups and compare both economic and clinical benefits among different indication. By comparing economic and clinical benefits of remote monitoring by different subgroups, the investigators might be able to set a guideline on which group of patients should be strongly suggested for remote monitoring utilization.

Therefore, the investigators perform a prospective study in Korean population to compare economic and clinical benefits of RM compared to conventional follow-up in overall study cohort and by different subgroups. (ICD & CRT-D).

DETAILED DESCRIPTION:
The investigators propose to prospectively recruit 556 patients with ICD or CRT-D implantation in 10 sites in Korea.

* Eligible patients should be enrolled in remote monitoring system 0 to 45 days after successful device implantation and then randomly assigned in a 1:1 ratio to the RM or conventional follow-up group.
* In the RM follow-up arm, the patients are not mandated to visit the clinic unless there is unscheduled call due to adverse event notification.
* In the conventional follow-up arm, the patients should be seen at the clinic according to each center's custom but no longer than 1 year between each visit. Follow-up should be continued accordingly until two-years of device implant.

ELIGIBILITY:
Inclusion Criteria:

1. All ICD and CRT-D patients who are over the age of 18
2. Ability to provide informed consent and to complete the study and required follow-up

Exclusion Criteria:

1. Those who refuse to participate in the trial.
2. Those who refuse to use remote monitoring system or who live in an environment where remote monitoring system cannot be utilized.
3. Patient who refuse to use or expected to use less than 75% of remote monitoring system.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1140 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse event | up to 2 years
  Definition of major adverse events (MAE)
  1. fatal or life-threatening
  2. prompted or prolonged a hospitalization;
  3. caused major or permanent disability or injury;
  4. required an intervention to prevent permanent disability or injury
Major adverse event, including death from any cause, cardiovascular, and procedure- or device-related MAE. | up to 2 years
  Definition of device-related adverse events
  1. delivery of ≥1 inappropriate shock(s);
  2. delivery of ≥2 symptomatic inappropriate ATP;
  3. symptomatic defibrillator-mediated tachycardia;
  4. infection or extrusion of the ICD;
  5. ineffective pacing;
  6. intermittent or permanent undersensing;
  7. clinical phrenic stimulation; and
  8. lead or pulse generator dysfunction.

SECONDARY OUTCOMES:
Economic benefit by remote monitoring | up to 2 years
  - Cost Incurred by the patient towards the transportation
Economic benefit by remote monitoring | up to 2 years
  - Consultation fee
Economic benefit by remote monitoring | up to 2 years
  - Patient Travel Time
Economic benefit by remote monitoring | up to 2 years
  - Patient consultation Time
Economic benefit by remote monitoring | up to 2 years
  - Administrative activities Time
Economic benefit by remote monitoring | up to 2 years
  - Device interrogation Time
Economic benefit by remotemonitoring | up to 2 years
  - Cost towards loss of employment for time spent in hospital for check-up of patient
Economic benefit by remotemonitoring | up to 2 years
  - Cost towards loss of employment of attendant for time spent in hospital for check-up of patient (dependent)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No